CLINICAL TRIAL: NCT03179670
Title: Interest of a Systematic Assessment of the Treatment of Lower Urinary Tract Symptoms (LUTS) in the Management of Benign Prostatic Hyperplasia (BPH) in Urology
Brief Title: Interest of a Systematic Assessment of the Treatment of LUTS in the Management of BPH
Acronym: UROEVAL
Status: Completed | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Collaborators: ClinSearch (Other)
Responsible Party: Sponsor
Other Study IDs: KMD 3213-FR-NIS-0019
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The high level of unsatisfactory outcome observed in patients treated for LUTS associated with BPH with respect to the different existing therapeutic options strongly emphasizes the need for treatment optimisation in daily practice by a careful LUTS monitoring and treatment adjustment when needed. The poorer outcome observed in patients for whom treatment has been initiated recently suggests that the duration of the disease itself may influence the patient satisfaction.To achieve this goal, we propose to systematically assess LUTS associated with BPH in patients treated for at least 6 months and to assess whether an alpha-blocker therapy initiation/modification may improve the outcome in case of persisting symptoms. We also investigate the influence of the symptom duration on the frequency of unsatisfactory outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 60 years or more suffering from LUTS/BPH AND medically treated for at least 6 months.

Exclusion Criteria:

* Patients with prostate cancer
* Patients requiring surgical treatment
* The absence of Lower Urinary Tract Symptoms
* Treatment initiation for less than 6 months
* Cognitive disorders or other pathologies leading to the inability to give its consent to the collection of data.
* Refusal to participate.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The frequency of patients with IPSS score <8 after three months of treatment with alpha-blockers is about 40%. The sample size required to detect a proportion of 40% with a precision of 0.04 is 550 patients. Based on a literature review of Lacoin et al, the frequency of treated patients with LUTS associated with BPH with an IPSS ≥ 8 is approximately 60%. Thus, 917 patients will be needed to obtain a sample of 550 patients with treatment of alpha-blockers (550/0.6 = 917).
  Considering 10% of patients lost for follow-up or refusing treatment change, the total number required is estimated at about 1,000 patients.
Sampling Method: Probability Sample
Enrollment: 625 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients treated for LUTS associated with BPH displaying unsatisfactory outcome after at least 6 months of treatment and not requiring surgical treatment. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- LBR, Puteaux, France

IPD SHARING:
Plan to Share IPD: No